CLINICAL TRIAL: NCT04357873
Title: Phase II Basket Trial Evaluating the Efficacy of a Combination of Pembrolizumab and Vorinostat in Patients With Recurrent and/or Metastatic Squamous Cell Carcinoma
Brief Title: Efficacy of Immunotherapy Plus a Drug in Patients With Progressive Advanced Mucosal Cancer of Different Locations
Acronym: PEVOsq
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Fondation ARC (Other); ERA-NET (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-GMP-1908; 2019-003839-33 (EudraCT Number)
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-02

CONDITIONS: Squamous Cell Lung Cancer; Vulvar Cancer; Penile Cancer; Cervix Cancer; Head and Neck Squamous Cell Carcinoma; Anal Cancer
Keywords: squamous cell carcinoma; squamous cell cancer
MeSH Terms: conditions — Vulvar Neoplasms; Penile Neoplasms; Uterine Cervical Neoplasms; Squamous Cell Carcinoma of Head and Neck; Anus Neoplasms; Carcinoma, Squamous Cell; Neoplasms, Squamous Cell | interventions — pembrolizumab; Vorinostat

STUDY DESIGN:
Intervention Model Description: 6 independent cohorts (head and neck, cervix, lung, anus, vulva, and penis) evaluating the association of pembrolizumab and vorinostat
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- pembrolizumab + vorinostat (Experimental): Pembrolizumab: 200 mg every 3 weeks, up to 35 administrations
  Vorinostat: 400 mg once daily, until progression
  Interventions: Drug: pembrolizumab; vorinostat

INTERVENTIONS:
Drug: pembrolizumab; vorinostat — Pembrolizumab: 200 mg every 3 weeks, up to 35 administrations
  Vorinostat: 400 mg once daily, until progression
  Other Names: KEYTRUDA; ZOLINZA

SUMMARY:
Interventional study evaluating the efficacy of an immunotherapy (pembrolizumab) in combination with a targeted therapy (vorinostat) in patient with recurrent and/or metastatic squamous cell carcinoma (localisations : head and neck, lung, cervix, anus, vulva, and penis)

DETAILED DESCRIPTION:
Open-label, non-randomized, multi-center, basket phase II trial, evaluating the efficacy of pembrolizumab in combination with vorinostat in adult patients with recurrent and/or metastatic squamous cell carcinoma of different locations.

Antitumor activity of the combination will be evaluated using the objective response rate (ORR) during treatment (investigator assessment).

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years old.
2. Patients with Eastern Cooperative Oncology Group (ECOG) performance status ≤1.
3. Patients must have histologically confirmed recurrent and/or metastatic squamous cell carcinoma of the head and neck, cervix, lung, anus, vulva, or penis.
4. Patients must have radiologically confirmed progressive recurrent and/or metastatic disease.
5. Patients naive or previously treated for recurrent and/or metastatic disease for which a treatment with an anti-PD1/PD-L1 agents and vorinostat is an acceptable option according to investigator.
6. Disease amenable to biopsy for study purpose.
7. Measurable disease according to RECIST v1.1.
8. Adequate renal function: serum creatinine ≤1.5 x upper limit of normal (ULN) (OR creatinine clearance [Cockcroft and Gault] ≥30 mL/min for participant with creatinine levels >1.5 × ULN) within 14 days prior inclusion.
9. Adequate liver function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤3 × ULN (≤5 ULN when documented liver metastases) and total bilirubin level ≤1.5 × ULN, within 14 days prior inclusion.
10. Adequate bone marrow function: absolute neutrophil count (ANC) ≥1,000/mm³, platelet count ≥100,000/mm³, and hemoglobin ≥9 g/dL, within 14 days prior inclusion.
11. Adequate coagulation: prothrombin time (PT)/international normalized ratio (INR) ≤1.5 × ULN within 14 days prior inclusion If participant is receiving anticoagulant therapy then the PT or activated partial thromboplastin time (aPTT) should be within the therapeutic range of intended use of anticoagulant.
12. Female of child-bearing potential must have a negative serum pregnancy test within 72 h before starting study treatment.
13. Female of childbearing potential, must use "highly effective" methods of contraception for the study duration and for 4 months following the last dose of pembrolizumab and 6 months following the last dose of vorinostat.
14. Male participants must agree to use an effective contraceptive for the duration of the trial and for at least 4 months after the last the last dose of pembrolizumab and 6 months following the last dose of vorinostat (to allow for effective elimination of the study drugs). Also, they should refrain from donating sperm during this period.
15. Patients must be willing and able to comply with the protocol for the duration of the study including scheduled visits, treatment plan, and laboratory tests.
16. Patients must be willing and able to comply with other study procedures, including a baseline tumor biopsy and a series of blood samples throughout the study.
17. Patients able to swallow oral medications.
18. Patients must be affiliated to a Social Security System (or equivalent).
19. Patients must have signed a written informed consent prior to any trial-specific procedures. When the patient is physically unable to give their written consent, a trusted person of their choice, independent from the investigator or the sponsor, can confirm in writing the patient's consent.

Exclusion Criteria:

1. Prior treatment with anti-PD-1/PD-L1 agents or histone deacetylases (HDAC) inhibitors.
2. Patients with central nervous system involvement that has not been controlled for >3 months.
3. Patients with no other site for biopsy than bone lesions.
4. Patients with other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study, including uncontrolled diabetes, cardiac disease, uncontrolled hypertension, congestive cardiac failure, ventricular arrhythmias, active ischemic heart disease, myocardial infection within one year, chronic liver or renal disease, active gastrointestinal tract ulceration, severely impaired lung function.
5. Known history of human immunodeficiency virus (HIV), Hepatitis B virus (HBV; defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (HCV; defined as HCV RNA detected) virus infection.
6. History of autoimmune disease with the exception of:

   * (1) Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone,
   * (2) Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen,
   * (3) Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) provided that they meet the following conditions: (i) Rash must cover less than 10% of body surface area; (ii) Disease is well controlled at baseline and only requiring low potency topical steroids; (iii) No acute exacerbations of underlying condition within the previous 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoid, biologic agents, oral calcineurin inhibitors, high-potency or oral steroids).
7. History of allogeneic organ or bone marrow transplantation.
8. History of non-infectious pneumonitis that required steroids or has current pneumonitis.
9. Has an active infection requiring systemic therapy.
10. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
11. Known prior severe hypersensitivity to investigational products or its excipients,
12. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks [could consider shorter interval for kinase inhibitors or other short half-life drugs] prior to first dose of study treatments.

    Note: Participants must have recovered from all adverse events due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible.
13. Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system disease.
14. Major surgery within 28 days prior to the first dose of study treatments. Note: Local surgery of isolated lesions for palliative intent is acceptable.
15. Current or prior use of immunosuppressive medication within 7 days before the first dose of pembrolizumab. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection),
    * Systemic corticosteroids at physiologic doses ≤10 mg/day of prednisone or its equivalent,
    * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
16. Patients using drugs that could have pharmacokinetics interaction with investigational drugs. This includes, but is not limited to, valproic acid, coumarin-derivative anticoagulants, drugs that disrupt electrolyte levels, drugs that may prolong QT.
17. Pregnant women or women who are breast-feeding.
18. Patients enrolled in another therapeutic study within 30 days prior to inclusion and during the treatment period. Patients can participate in an independent approved non-interventional studies.
19. Patients unwilling or unable to comply with the medical follow-up required by the trial because of geographic, familial, social, or psychological reasons.
20. Persons deprived of their liberty or under protective custody or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR), investigator assessment | From inclusion to first and subsequent tumor assesment or progression, up to 24 months
  Investigators will assess the ORR. The ORR is defined in each cohort as the percentage of evaluable patients for ORR, designate as the proportion of patients with best response of complete response (CR) or a partial response (PR) during treatment according to response evaluation criteria in solid tumors version 1.1 (RECIST v1.1).

SECONDARY OUTCOMES:
Objective Response Rate (ORR), central assessment | From inclusion to first and subsequent tumor assesment or progression, up to 36 months
  ORR defined as the proportion of patients with best response of CR or PR during treatment, as assessed by a central radiological panel according to RECIST v1.1.
immune Objective Response Rate (iORR), central assessment | From inclusion to first and subsequent tumor assesment or progression, up to 36 months
  ORR defined as the proportion of patients with best response of CR or PR during treatment, as assessed by a central radiological panel according to immune-specific response criteria.
Duration Of Response (DOR) | From the first assessment of a CR or PR until the date of the first occurrence of PD or death from any cause
  DOR will be evaluated in patients with either CR or PR. DOR is defined as the time from the first assessment of a CR or PR until the date of the first occurrence of progressive disease (PD) or death from any cause (if death occurred within predefined period), whichever occurs first.
Progression Free Survival (PFS) | From inclusion to disease progression or death, up to 36 months
  PFS is defined per RECIST v1.1 as the time from inclusion until disease progression (per RECIST v1.1) or death from any cause, whichever occurs first. At the time of analysis, a patient alive and without disease progression will be censored at the date of the last tumor assessment. Patients alive without disease progression who started a new anticancer therapy will be censored at the date of the last tumor assessment prior to the start of the new anticancer therapy.
immune Progression Free Survival (iPFS) | From inclusion to disease progression or death, up to 36 months
  iPFS is defined per immune-specific response evaluation criteria in solid tumors (iRECIST) as the time from inclusion until confirmed disease progression (per iRECIST), or death from any cause, whichever occurs first. At the time of analysis, a patient alive and without progression will be censored at the date of the last tumor assessment. Patients alive without disease progression who started a new anti-cancer therapy will be censored at the date of the last tumor assessment prior to the start of the new anticancer therapy.
Overall Survival (OS) | From inclusion to death from any cause, up to 36 months
  OS is defined as the time from inclusion until death from any cause. Patients who are alive at last follow-up news will be censored at this date.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Le Tourneau, MD, Principal Investigator — Institut Curie
Locations (14):
- France (14):
  - Institut de Cancérologie de l'Ouest - Site Paul Papin, Angers
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre George François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut de Cancérologie de Lorraine, Nancy
  - Institut de Cancérologie de l'Ouest (site René Gauducheau), Nantes
  - Institut Curie, Paris
  - Centre Hospitalier Lyon Sud - Hospices Civils de Lyon, Pierre-Bénite
  - Institut Godinot, Reims
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, Toulouse

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.

REFERENCES:
- [Derived] Filippini DM, Cabarrou B, Dupain C, Halladjian M, Coquan E, Sablin MP, Mazzarella L, Francisco M, Servant N, Tonini MM, Hundt AF, Castel-Ajgal Z, You B, Bigot F, Ghiringhelli F, Vansteene D, Gomez-Roca C, Cousin S, Lambert A, Saada-Bouzid E, Durando X, Abdeddaim C, Borel C, Chaltiel R, Borcoman E, Legrand F, Bernhart S, Jimenez M, Bieche I, Filleron T, Le Tourneau C, Kamal M, Jeannot E. HPV circulating tumor DNA to monitor response to pembrolizumab and vorinostat combination in patients with advanced HPV-related squamous-cell carcinomas. ESMO Open. 2026 Jan;11(1):106024. doi: 10.1016/j.esmoop.2025.106024. Epub 2025 Dec 29. PMID 41468684
- [Derived] Borcoman E, Cabarrou B, Francisco M, Bigot F, Ghiringhelli F, Vansteene D, Legrand F, Halladjian M, Dupain C, Le Saux O, Coutzac C, Borel C, Chaltiel R, You B, Gomez-Roca C, Cousin S, Coquan E, Lambert A, Saada-Bouzid E, Durando X, Saint-Ghislain M, Frige G, Guerini-Rocco E, Tonini MM, Bieche I, Castel-Ajgal Z, Marret G, Sablin MP, Jeannot E, Andre F, Filleron T, Jimenez M, Mazzarella L, Servant N, Kamal M, Le Tourneau C. Efficacy of pembrolizumab and vorinostat combination in patients with recurrent and/or metastatic squamous cell carcinomas: a phase 2 basket trial. Nat Cancer. 2025 Aug;6(8):1370-1383. doi: 10.1038/s43018-025-01004-2. Epub 2025 Jun 30. PMID 40588522

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/73/NCT04357873/Prot_SAP_000.pdf